CLINICAL TRIAL: NCT03285490
Title: A Phase 3, Double-Blind, Vehicle-Controlled, Randomized, Parallel Group, Multicenter, Efficacy and Safety Study of KX2-391 Ointment 1% in Adult Subjects With Actinic Keratosis on the Face or Scalp
Brief Title: A Multi-Center Study to Evaluate the Efficacy and Safety of KX2-391 Ointment 1% on Actinic Keratosis on Face or Scalp (AK004)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Almirall, S.A. (Industry)
Collaborators: Athenex, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KX01-AK-004; U1111-1191-8287 (Other: UTN)
Record Dates: First submitted 2017-09-07; First posted 2017-09-18 (Actual); Results first posted 2021-03-10 (Actual); Last update posted 2021-03-10 (Actual); Status verified 2021-02

CONDITIONS: Actinic Keratosis
Keywords: Actinic Keratosis; Keratosis; Keratosis, Actinic; Precancerous Conditions; Neoplasms; Sun Damaged Skin; Actinic Keratoses
MeSH Terms: conditions — Keratosis, Actinic; Keratosis; Precancerous Conditions; Neoplasms

STUDY DESIGN:
Intervention Model Description: This study tested KX2-391 Ointment 1% against a placebo.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All Central Vendors and the sponsor were masked. The sponsor was unblind at the end of Day 57.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- KX2-391 Ointment 1% (Experimental): KX2-391 Ointment was applied once daily for 5 consecutive days on the face or scalp.
  Interventions: Drug: KX2-391 Ointment 1%
- Placebo (Placebo Comparator): The Vehicle Ointment was applied once daily for 5 consecutive days on the face or scalp.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: KX2-391 Ointment 1% — Dose: 1% (250 mg single-use packets); Dosage form: Ointment; Route of administration: Topical
  Arms: KX2-391 Ointment 1%
Drug: Placebo — Dosage form: Ointment; Route of administration: Topical
  Arms: Placebo

SUMMARY:
This Phase III study was designed to evaluate the efficacy and safety of KX2-391 Ointment 1% in adult participants when applied to an area of skin containing 4-8 stable, clinically typical actinic keratosis (AK) lesions on the face or scalp.

DETAILED DESCRIPTION:
This study was a double-blinded, multicenter, efficacy, and safety study of KX2-391 ointment administered topically to the face or scalp of participants with AK.

The study consisted of Screening, Treatment, Follow-up, and Recurrence Follow-up Periods. Eligible participants received up to 5 consecutive days of topical treatment. Efficacy (lesion counts) and safety evaluations were performed.

ELIGIBILITY:
Inclusion Criteria

1. Males and females greater than or equal to (>=) 18 years old.
2. A defined area on the face or scalp contains 4 to 8 clinically typical, visible, and discrete AK lesions.
3. Participants who in the judgment of the Investigator, were in good general health.
4. Females were postmenopausal (greater than [>] 45 years of age with at least 12 months of amenorrhea), surgically sterile (by hysterectomy, bilateral oophorectomy, or tubal ligation); or, if of childbearing potential, were using highly effective contraception for at least 30 days or 1 menstrual cycle, whichever was longer, prior to study treatment and agreed to continue to use highly effective contraception for at least 30 days following their last dose of study treatment. Highly effective contraception includes oral hormonal contraceptives, hormonal contraceptive implant, injection or patch, intrauterine device or complete abstinence from sexual intercourse.
5. Sexually active males who had not had a vasectomy, and whose partner was reproductively capable, must had agreed to use barrier contraception from Screening through 90 days after their last dose of study treatment.
6. All participants must had agreed not to donate sperm or eggs or attempt conception from Screening through 90 days following their last dose of study treatment.
7. Willing to avoid excessive sun or ultraviolet exposure.
8. Able to comprehend and were willing to sign the informed consent form (ICF).

Exclusion Criteria

1. Clinically atypical and/or rapidly changing AK lesions on the treatment area.
2. Location of the selected area is:

   * On any location other than the face or scalp.
   * Within 5 centimeters (cm) of an incompletely healed wound.
   * Within 5 cm of a suspected basal cell carcinoma (BCC) or squamous cell carcinoma (SCC).
3. Been previously treated with KX2-391 Ointment.
4. Anticipated need for in-patient hospitalization or in-patient surgery from Day 1 to Day 57.
5. Treatment with 5-fluorouracil (5-FU), imiquimod, ingenol mebutate, diclofenac, photodynamic therapy, or other treatments for AK within the treatment area or within 2 cm of the treatment area, within 8 weeks prior to the Screening visit.
6. Use of the following therapies and/or medications within 2 weeks prior to the Screening visit:

   * Cosmetic or therapeutic procedures (e.g., use of liquid nitrogen, surgical excision, curettage, dermabrasion, medium or greater depth chemical peel, laser resurfacing) within the treatment area or within 2 cm of the selected treatment area.
   * Acid-containing therapeutic products (eg, salicylic acid or fruit acids, such as alpha- and beta-hydroxyl acids and glycolic acids), topical retinoids, or light chemical peels within the treatment area or within 2 cm of the selected treatment area.
   * Topical salves (non-medicated/non-irritant lotion and cream were acceptable) or topical steroids within the treatment area or within 2 cm of the selected treatment area; artificial tanners within the treatment area or within 5 cm of the selected treatment area.
7. Use of the following therapies and/or medications within 4 weeks prior to the Screening visit:

   * Treatment with immunomodulators (eg, azathioprine), cytotoxic drugs (eg, cyclophosphamide, vinblastine, chlorambucil, methotrexate) or interferons/interferon inducers.
   * Treatment with systemic medications that suppress the immune system (eg, cyclosporine, prednisone, methotrexate, alefacept, infliximab).
8. Use of systemic retinoids (eg, isotretinoin, acitretin, bexarotene) within 6 months prior to the Screening visit.
9. A history of sensitivity and/or allergy to any of the ingredients in the study medication.
10. A skin disease (e.g., atopic dermatitis, psoriasis, eczema) or condition (e.g., scarring, open wounds) that, in the opinion of the Investigator, might interfere with the study conduct or evaluations, or which exposes the participant to unacceptable risk by study participation.
11. Other significant uncontrolled or unstable medical diseases or conditions that, in the opinion of the Investigator, would expose the participant to unacceptable risk by study participation.
12. Females who were pregnant or nursing.
13. Participated in an investigational drug trial during which an investigational study medication was administered within 30 days or 5 half-lives of the investigational product, whichever was longer, before dosing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 351 (Actual)
Dates: Start 2017-09-15 (Actual); Primary Completion 2018-05-07 (Actual); Study Completion 2019-04-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jane Fang, MD, Study Chair — Athenex, Inc.
Locations (30):
- United States (30):
  - Alliance Dermatology, Phoenix, Arizona
  - Synexus US, Tucson, Arizona
  - Burke Pharmaceutical Research, Hot Springs, Arkansas
  - Dermatology Specialists, Inc., Murrieta, California
  - Dermatology Specialists, Inc., Oceanside, California
  - Skin Surgery Medical Group, Inc., San Diego, California
  - Synexus, Santa Rosa, California
  - AboutSkin Dermatology, Greenwood Village, Colorado
  - Study Protocol, Inc, Boynton Beach, Florida
  - Sweet Hope Research Specialty, Inc., Miami Lakes, Florida
  - Forward Clinical Trials, Inc., Tampa, Florida
  - Laser & Skin Surgery Center of Indiana, Carmel, Indiana
  - Dawes Fretzin Clinical Research Group, Indianapolis, Indiana
  - DS Research, Louisville, Kentucky
  - Clinical Trials of SWLA, LLC, Lake Charles, Louisiana
  - Hamzavi Dermatology, Fort Gratiot, Michigan
  - Medisearch Clinical Trials, Saint Joseph, Missouri
  - Henderson Dermatology Research, Henderson, Nevada
  - Activmed Practices & Research, Inc, Portsmouth, New Hampshire
  - Union Square Laser Dermatology, New York, New York
  - Aventiv Research Inc., Dublin, Ohio
  - Oregon Medical Research Center, Portland, Oregon
  - Clinical Research Center of the Carolinas, Charleston, South Carolina
  - Dermatology Associates Of Knoxville, PC, Knoxville, Tennessee
  - Rivergate Dermatology Clinical Research, Springfield, Tennessee
  - DermResearch, Austin, Texas
  - Suzanne Bruce and Associates, P.A., The Center for Skin Research, Houston, Texas
  - Clinical Trials of Texas, Inc., San Antonio, Texas
  - The Education & Research Foundation, Inc., Lynchburg, Virginia
  - Dermatology Associates of Seattle, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Blauvelt A, Kempers S, Lain E, Schlesinger T, Tyring S, Forman S, Ablon G, Martin G, Wang H, Cutler DL, Fang J, Kwan MR; Phase 3 Tirbanibulin for Actinic Keratosis Group. Phase 3 Trials of Tirbanibulin Ointment for Actinic Keratosis. N Engl J Med. 2021 Feb 11;384(6):512-520. doi: 10.1056/NEJMoa2024040. PMID 33567191

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 31 sites in the United States between 15-September-2017 to 24-April-2019.
Pre-assignment Details: A total of 410 participants were screened, of which 351 participants were enrolled, 173 were randomized to vehicle control (118 face, 55 scalp) and 178 to KX2-391 ointment 1 percent (%) (119 face, 59 scalp). This study consisted of 2 periods i.e., Treatment and response assessment period (Baseline up to Day 57) followed by Recurrence follow-up period (12 months post-Day 57).
Groups:
- Placebo: Vehicle Ointment was applied topically once daily for 5 consecutive days in a treatment area of 25 centimeter square (cm^2) on face or scalp.
- KX2-391 Ointment 1%: KX2-391 Ointment 1% was applied topically once daily for 5 consecutive days in a treatment area of 25 cm^2 on face or scalp.
Period: Treatment and Response Assessment Period
Arm/Group | Placebo | KX2-391 Ointment 1%
Started | 173 | 178
Completed | 173 | 178
Not Completed | 0 | 0
Period: Recurrence Follow-up Period
Arm/Group | Placebo | KX2-391 Ointment 1%
Started (Number of participants who achieved 100% AK clearance at Day 57 visit had entered the recurrence follow-up period.) | 22 | 97
Completed | 4 | 36
Not Completed | 18 | 61
Not completed — Withdrawal by Subject | 0 | 1
Not completed — AK recurrence during Recurrence Follow-Up Period | 18 | 60

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population included all randomized participants.
Groups:
- Placebo: Vehicle Ointment was applied topically once daily for 5 consecutive days in a treatment area of 25 cm^2 on face or scalp.
- Total: Total of all reporting groups
Arm/Group | Placebo | KX2-391 Ointment 1% | Total
Number analyzed (Participants) | 173 | 178 | 351
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.2 (8.86) | 69.1 (8.69) | 69.7 (8.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 20 | 43
  Male | 150 | 158 | 308
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 11 | 19
  Not Hispanic or Latino | 165 | 167 | 332
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 173 | 177 | 350
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Number of AK lesions at baseline [Mean (Standard Deviation); unit: lesions] | 5.8 (1.20) | 6.0 (1.27) | 5.9 (1.24)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Complete (100%) Clearance of Actinic Keratosis (AK) Lesions
Description: Complete clearance rate was defined as the percentage of participants at Day 57 with no clinically visible AK lesions in the treatment area.
Time Frame: Day 57
Population: ITT population included all randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | KX2-391 Ointment 1%
Number analyzed (Participants) | 173 | 178
percentage of participants | 13 | 54
Statistical Analysis 1: Comparison: Placebo vs KX2-391 Ointment 1%; Statistical significance in the study for Day 57 complete clearance rate was analyzed using a Cochran-Mantel-Haenszel model controlling for treatment location (face or scalp) and treatment group (Placebo versus KX2-391 Ointment 1%); Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — P-value threshold for statistical significance was 0.5%

2. Secondary Outcome: Percentage of Participants With Partial Clearance Rate of Actinic Keratosis Lesions at Day 57
Description: Partial clearance rate of AK lesions was defined as the percentage of participants with a greater than or equal to (>=) 75% reduction in the number of AK lesions identified at Baseline (Day 1 predose) in the treatment area.
Time Frame: Day 57
Population: ITT population included all randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | KX2-391 Ointment 1%
Number analyzed (Participants) | 173 | 178
percentage of participants | 20 | 76
Statistical Analysis 1: Comparison: Placebo vs KX2-391 Ointment 1%; Statistical significance in the study for Day 57 partial clearance rate was analyzed using a Cochran-Mantel-Haenszel model controlling for treatment location (face or scalp) and treatment group (Placebo versus KX2-391 Ointment 1%); Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — P-value threshold for statistical significance was 0.5%

3. Secondary Outcome: Overall Change From Baseline in Actinic Keratosis Lesion Counts at Days 8, 15, 29 and 57
Description: Overall the change from baseline in lesion count at each visit were summarized and reported using descriptive statistics by treatment location (face or scalp).
Time Frame: Days 8, 15, 29 and 57
Population: ITT population included all randomized participants.
Measure: Median (Full Range); unit: lesion count
Arm/Group | Placebo | KX2-391 Ointment 1%
Number analyzed (Participants) | 173 | 178
lesion count
  Day 8: number analyzed (Participants) | 170 | 159
  Day 8 | 0.0 [-8 to 1] | -1.0 [-7 to 3]
  Day 15: number analyzed (Participants) | 173 | 169
  Day 15 | -1.0 [-7 to 1] | -4.0 [-8 to 3]
  Day 29: number analyzed (Participants) | 172 | 177
  Day 29 | -1.0 [-7 to 2] | -5.0 [-8 to 1]
  Day 57 | -1.0 [-8 to 2] | -5.0 [-8 to 1]

4. Secondary Outcome: Percentage of Participants With Recurrence of Actinic Keratosis Lesions Who Achieved Complete Clearance at Day 57
Description: Recurrence rate was estimated based on Kaplan-Meier method, with recurrence define as appearance of any AK lesions in the treatment area, including those recurred or newly identified.
Time Frame: 3, 6, 9 and 12 months post-Day 57
Population: Recurrence follow-up population included all participants in the ITT Population who achieved complete clearance at the Day 57 visit. The recurrence rate was evaluated only for KX2-391 Ointment 1% arm, pre-specified in protocol.
Measure: Number; unit: percentage of participants
Arm/Group | KX2-391 Ointment 1%
Number analyzed (Participants) | 96
percentage of participants
  3 months post-Day 57 | 27
  6 months post-Day 57: number analyzed (Participants) | 70
  6 months post-Day 57 | 31
  9 months post-Day 57: number analyzed (Participants) | 48
  9 months post-Day 57 | 27
  12 months post-Day 57: number analyzed (Participants) | 35
  12 months post-Day 57 | 23

5. Secondary Outcome: Number of Participants With Maximal Post Baseline Local Skin Reaction (LSR)
Description: Maximal post baseline LSR was defined as the highest grade of any LSR reported at any post baseline visits for a participant. The LSR assessment was an Investigator's (or sub-investigator's) assessment of the following signs on the treatment area: erythema, flaking/scaling, crusting, swelling, vesiculation/pustulation, and erosion/ulceration. The LSRs were graded on a 4-point scale ranging from 0=absent, 1=mild (slightly, barely perceptible), 2=moderate (distinct presence), and 3=severe (marked, intense).
Time Frame: Day 57
Population: Safety analysis set included participants who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | KX2-391 Ointment 1%
Number analyzed (Participants) | 173 | 178
Participants
  Erythema-Grade 0 | 79 | 3
  Erythema-Grade 1 | 81 | 47
  Erythema-Grade 2 | 13 | 111
  Erythema-Grade 3 | 0 | 17
  Flaking/Scaling-Grade 0 | 82 | 8
  Flaking/Scaling-Grade 1 | 69 | 60
  Flaking/Scaling-Grade 2 | 21 | 90
  Flaking/Scaling-Grade 3 | 1 | 20
  Crusting-Grade 0 | 148 | 92
  Crusting-Grade 1 | 19 | 51
  Crusting-Grade 2 | 6 | 30
  Crusting-Grade 3 | 0 | 5
  Swelling-Grade 0 | 169 | 110
  Swelling-Grade 1 | 4 | 47
  Swelling-Grade 2 | 0 | 20
  Swelling-Grade 3 | 0 | 1
  Vesiculation/Pustulation-Grade 0 | 172 | 166
  Vesiculation/Pustulation-Grade 1 | 1 | 11
  Vesiculation/Pustulation-Grade 2 | 0 | 0
  Vesiculation/Pustulation-Grade 3 | 0 | 1
  Erosion/Ulceration-Grade 0 | 171 | 156
  Erosion/Ulceration-Grade 1 | 2 | 18
  Erosion/Ulceration-Grade 2 | 0 | 4
  Erosion/Ulceration-Grade 3 | 0 | 0

6. Secondary Outcome: Number of Participants With Pigmentation and Scarring in the Treatment Area
Description: Absence or presence of pigmentation (i.e., hypopigmentation and hyperpigmentation) and scarring in the treatment area were assessed.
Time Frame: Baseline (Day 1 predose), Days 5, 8, 15, 29 and 57
Population: Safety Population included all randomized participants who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | KX2-391 Ointment 1%
Number analyzed (Participants) | 173 | 178
Participants
  Hypopigmentation: Baseline | 26 | 30
  Hypopigmentation: Day 5 | 26 | 28
  Hypopigmentation: Day 8 | 23 | 30
  Hypopigmentation: Day 15 | 21 | 31
  Hypopigmentation: Day 29 | 21 | 32
  Hypopigmentation: Day 57 | 21 | 29
  Hyperpigmentation: Baseline | 33 | 36
  Hyperpigmentation: Day 5 | 30 | 33
  Hyperpigmentation: Day 8 | 30 | 34
  Hyperpigmentation: Day 15 | 27 | 32
  Hyperpigmentation: Day 29 | 24 | 29
  Hyperpigmentation: Day 57 | 25 | 25
  Scarring: Baseline | 9 | 11
  Scarring: Day 5 | 8 | 13
  Scarring: Day 8 | 8 | 11
  Scarring: Day 15 | 9 | 9
  Scarring: Day 29 | 8 | 9
  Scarring: Day 57 | 10 | 9

7. Secondary Outcome: Number of Participants With Adverse Event (AE), Treatment-emergent Adverse Events (TEAEs), Serious Adverse Events (SAEs), Events of Special Interests
Description: An AE was defined as any untoward medical occurrence in participant which does not necessarily have causal relationship with treatment. An AE was any unfavorable and unintended sign (including abnormal laboratory finding), symptom, or disease temporally associated with use of medicinal product, whether or not considered related to medicinal product. An SAE was any untoward medical occurrence that at any dose resulted in death; was life threatening; required persistent/significant disability/incapacity; resulted in initial or prolonged in patient hospitalization; was congenital anomaly/birth defect or otherwise considered medically important. TEAEs (serious and non-serious) were defined as either those AEs with onset after first dose or those pre-existing AEs that worsen after first dose. Events of special interest included skin cancers (including basal cell carcinoma, squamous cell carcinoma, melanoma and their location and treatment area), ocular exposure, overdose, and pregnancy.
Time Frame: Baseline (Day 1 predose) up to Day 57
Population: Safety Population included all randomized participants who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | KX2-391 Ointment 1%
Number analyzed (Participants) | 173 | 178
Participants
  Participants with AE | 73 | 71
  Participants with any TEAE | 67 | 67
  Participants with any SAE | 4 | 1
  Participants with events of special interest | 4 | 4

8. Secondary Outcome: Number of Participants With Adverse Events, Serious Adverse Events, Events of Special Interests Within the Treatment Area After Day 57 and up to 12 Months Post-Day 57
Description: An AE was defined as any untoward medical occurrence in participant which does not necessarily have causal relationship with treatment. An AE was any unfavorable and unintended sign (including abnormal laboratory finding), symptom, or disease temporally associated with use of medicinal product, whether or not considered related to medicinal product. An SAE was any untoward medical occurrence that at any dose resulted in death; was life threatening; required persistent/significant disability/incapacity; resulted in initial or prolonged in patient hospitalization; was congenital anomaly/birth defect or otherwise considered medically important. Events of special interest included skin cancers (including basal cell carcinoma, squamous cell carcinoma, melanoma and their location and treatment area), ocular exposure, overdose, and pregnancy.
Time Frame: From Day 57 up to 12-months post-Day 57
Population: Recurrence follow-up population included all participants in the ITT Population who achieved complete clearance at the Day 57 visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | KX2-391 Ointment 1%
Number analyzed (Participants) | 22 | 97
Participants
  Participants with any AE | 0 | 2
  Participants with any SAE | 0 | 0
  Participants with events of special interest | 1 | 0

9. Secondary Outcome: Number of Participants With Clinically Significant Safety Observations- Hematology, Blood Chemistry, Urinalysis
Description: Assessed laboratory parameters included hematology, blood chemistry and urinalysis. Clinical significance and abnormal observations were determined by the investigator.
Time Frame: From Baseline (Day 1 predose) up to Day 57
Population: Safety Population included all randomized participants who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | KX2-391 Ointment 1%
Number analyzed (Participants) | 173 | 178
Participants
  Hematology | 0 | 0
  Blood chemistry | 4 | 0
  Urinalysis | 0 | 1

10. Secondary Outcome: Number of Participants With Clinically Significant Safety Observations- Vital Signs
Description: Vital signs included measurement of pulse rate, systolic and diastolic blood pressure, respiratory rate, and body temperature. Clinical significance was determined by the investigator.
Time Frame: From Baseline (Day 1 predose) up to Day 57
Population: Safety Population included all randomized participants who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | KX2-391 Ointment 1%
Number analyzed (Participants) | 173 | 178
Participants | 0 | 0

11. Secondary Outcome: Number of Participants With Clinically Significant Safety Observations- Physical Examination
Description: A physical examination included weight and height measurements was performed. Clinical significance was determined by the investigator.
Time Frame: From Baseline (Day 1 predose) up to Day 57
Population: Safety Population included all randomized participants who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | KX2-391 Ointment 1%
Number analyzed (Participants) | 173 | 178
Participants | 0 | 0

12. Secondary Outcome: Number of Participants With Clinically Significant Safety Observations- Electrocardiograms (ECGs)
Description: ECG parameters included heart rhythm, heart rate, QRS intervals, QT intervals, RR intervals and corrected QT (QTc) intervals. Clinical significance was determined by the investigator.
Time Frame: From Baseline (Day 1 predose) up to Day 57
Population: Safety Population included all randomized participants who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | KX2-391 Ointment 1%
Number analyzed (Participants) | 173 | 178
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: From Baseline (Day 1 predose) up to 15 months (12 months post-Day 57)
Description: Safety population included all randomized participants who received at least one dose of study treatment.
Arm/Group | Placebo | KX2-391 Ointment 1%
All-Cause Mortality (participants affected / at risk) | 0/173 | 0/178
Serious Adverse Events (participants affected / at risk) | 4/173 | 1/178
Other Adverse Events (participants affected / at risk) | 72/173 | 72/178
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=173) | KX2-391 Ointment 1% (N=178)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Atrioventricular block complete (Cardiac disorders) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=173) | KX2-391 Ointment 1% (N=178)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Arrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Atrial flutter (Cardiac disorders) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Diplopia (Eye disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Bowel movement irregularity (Gastrointestinal disorders) | 1 (1) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Application site pruritus (General disorders) | 13 (13) | 19 (19)
Application site pain (General disorders) | 5 (5) | 24 (31)
Application site inflammation (General disorders) | 0 (0) | 1 (1)
Application site nodule (General disorders) | 0 (0) | 1 (1)
Application site paraesthesia (General disorders) | 1 (1) | 0 (0)
Application site scab (General disorders) | 0 (0) | 1 (1)
Chest discomfort (General disorders) | 0 (0) | 1 (1)
Influenza like illness (General disorders) | 1 (1) | 0 (0)
Nodule (General disorders) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1)
Peripheral swelling (General disorders) | 1 (1) | 0 (0)
Seasonal allergy (Immune system disorders) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 10 (10) | 8 (8)
Viral upper respiratory tract infection (Infections and infestations) | 4 (4) | 9 (9)
Cellulitis (Infections and infestations) | 1 (1) | 2 (2)
Sinusitis (Infections and infestations) | 3 (3) | 0 (0)
Urinary tract infection (Infections and infestations) | 3 (3) | 1 (1)
Influenza (Infections and infestations) | 2 (2) | 1 (1)
Angular cheilitis (Infections and infestations) | 0 (0) | 1 (1)
Application site folliculitis (Infections and infestations) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 1 (1)
Carbuncle (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0)
Herpes simplex (Infections and infestations) | 1 (1) | 0 (0)
Labyrinthitis (Infections and infestations) | 2 (2) | 0 (0)
Localised infection (Infections and infestations) | 1 (1) | 0 (0)
Onychomycosis (Infections and infestations) | 0 (0) | 1 (1)
Post procedural infection (Infections and infestations) | 0 (0) | 1 (1)
Postoperative wound infection (Infections and infestations) | 0 (0) | 1 (1)
Pyuria (Infections and infestations) | 0 (0) | 1 (1)
Streptococcal infection (Infections and infestations) | 1 (1) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 1 (1) | 0 (0)
Tooth infection (Infections and infestations) | 0 (0) | 1 (1)
Skin abrasion (Injury, poisoning and procedural complications) | 3 (4) | 4 (4)
Animal bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Face injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tooth fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 2 (2) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Blood testosterone decreased (Investigations) | 1 (1) | 0 (0)
Cardiac murmur (Investigations) | 0 (0) | 1 (1)
Crystal urine present (Investigations) | 0 (0) | 1 (1)
Prostatic specific antigen increased (Investigations) | 1 (1) | 0 (0)
Urobilinogen urine increased (Investigations) | 0 (0) | 1 (1)
Haemochromatosis (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (5) | 3 (3)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 3 (4)
Haemangioma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Renal cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Squamous cell carcinoma of head and neck (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 1 (1)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Nervous system disorder (Nervous system disorders) | 1 (1) | 0 (0)
Ketonuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (5)
Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Lentigo (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rosacea (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Scab (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Skin tightness (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Arthrodesis (Surgical and medical procedures) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 1 (1)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0)
Tongue disorder (Gastrointestinal disorders) | 0 (0) | 1 (1)
Bacteriuria (Infections and infestations) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Glycosuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Proteinuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Meniscus operation (Surgical and medical procedures) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2018-02-18): https://cdn.clinicaltrials.gov/large-docs/90/NCT03285490/Prot_000.pdf
  • Statistical Analysis Plan (2019-06-04): https://cdn.clinicaltrials.gov/large-docs/90/NCT03285490/SAP_001.pdf